CLINICAL TRIAL: NCT01768195
Title: Prophylactic Use of Entecavir for HBsAg Positive Lymphoma Patients Treated With Rituximab-based Immunochemotherapy
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking University (Other)
Responsible Party: Principal Investigator, Jun Zhu, Peking University Cancer Hospital & Institute, Peking University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PKU-2012111304
Record Dates: First submitted 2013-01-09; First posted 2013-01-15 (Estimated); Last update posted 2017-01-10 (Estimated); Status verified 2017-01

CONDITIONS: Hepatitis B
Keywords: Lymphoma; Hepatitis B Virus; Therapeutic Uses; Antiviral Agents; rituximab
MeSH Terms: conditions — Hepatitis B; Lymphoma | interventions — entecavir

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Entecavir prophylaxis (Experimental): Participants will initiate entecavir 0.5 mg/day orally on day 1 of the first course of immunochemotherapy and/or chemotherapy, and will be continued until 12 months after completion of the immunochemotherapy and/or chemotherapy.
  Interventions: Drug: Entecavir prophylaxis

INTERVENTIONS:
Drug: Entecavir prophylaxis — Entecavir 0.5mg daily from day 1 of immunochemotherapy and/or chemotherapy to 12 months after completing immunochemotherapy and/or chemotherapy.
  In patients with low load of hepatitis B virus DNA(≤2000 IU/ml), rituximab will be administrated at the beginning of entecavir prophylaxis. And in patients with high load of hepatitis B virus DNA(>2000 IU/ml), rituximab will be administrated when hepatitis B virus DNA decreased to the level of 2000 IU/ml after entecavir prophylaxis.
  Other Names: Baraclude

SUMMARY:
The purpose of this study is to identify the effect of prophylactic entecavir in HBsAg Positive lymphoma patients treated with rituximab-based immunochemotherapy.

DETAILED DESCRIPTION:
HBsAg Positive lymphoma patients are treated with entecavir when they receive rituximab-based immunochemotherapy. Entecavir 0.5mg daily is administrated from day 1 of immunochemotherapy and/or chemotherapy to 12 months after completing immunochemotherapy and/or chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* treatment-naive patients with B-cell lymphoma
* HBsAg positive at baseline
* treated with rituximab-based immunochemotherapy
* life expectancy of more than 3 months

Exclusion Criteria:

* younger than 18 years old
* HBsAg negative at baseline
* pregnant or lactating women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2013-01; Primary Completion 2017-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
the incidence of hepatitis B virus reactivation and hepatitis B virus reactivation related hepatitis | from the beginning of immunochemotherapy and/or chemotherapy to 24 months after the last cycle of immunochemotherapy and/or chemotherapy

SECONDARY OUTCOMES:
the incidence of hepatitis B virus virological response | from the beginning of immunochemotherapy and/or chemotherapy to 24 months after the last cycle of immunochemotherapy and/or chemotherapy
the incidence of hepatitis B virus serological response | from the beginning of immunochemotherapy and/or chemotherapy to 24 months after the last cycle of immunochemotherapy and/or chemotherapy
the incidence of hepatitis B virus maintained response | from the beginning of immunochemotherapy and/or chemotherapy to 24 months after the last cycle of immunochemotherapy and/or chemotherapy
the incidence of hepatitis B virus sustained response | from the beginning of immunochemotherapy and/or chemotherapy to 24 months after the last cycle of immunochemotherapy and/or chemotherapy
the incidence of hepatitis B virus relapse and relapse related hepatitis | from the beginning of immunochemotherapy and/or chemotherapy to 24 months after the last cycle of immunochemotherapy and/or chemotherapy

CONTACTS AND LOCATIONS:
Overall Officials: Jun Zhu, Principal Investigator — Peking University Cancer Hospital & Institute
Locations (13):
- China (13):
  - Peking University Cancer Hospital & Institute, Beijing, Beijing Municipality
  - 307 Hospital of the Chinese People's Liberation Army, Beijing, Beijing Municipality
  - 309 Hospital of the Chinese People's Liberation Army, Beijing, Beijing Municipality
  - Aerospace Central Hospital, Beijing, Beijing Municipality
  - Air Force General Hospital of the Chinese People's Liberation Army, Beijing, Beijing Municipality
  - Beijing Hospital, Beijing, Beijing Municipality
  - Cancer Institute & Hospital, Chinese Academy of Medical Sciences, Beijing, Beijing Municipality
  - First Hospital affiliated to General Hospital of the Chinese People's Liberation Army, Beijing, Beijing Municipality
  - General Hospital of Chinese People's Liberation Army, Beijing, Beijing Municipality
  - Peking Union Medical College Hospital, Beijing, Beijing Municipality
  - Peking University First Hospital, Beijing, Beijing Municipality
  - Peking University People's Hospital, Beijing, Beijing Municipality
  - Peking University Third Hospital, Beijing, Beijing Municipality